CLINICAL TRIAL: NCT06045481
Title: Postexposure Prophylaxis With Single Dose Doxycycline for the Prevention of Tick-borne Relapsing Fever
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2358-2023
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-05

CONDITIONS: Relapsing Fever, Tick-Borne
Keywords: Tick-borne Diseases; doxycycline; soldiers; israel defense forces medical corps
MeSH Terms: conditions — Relapsing Fever; Tick-Borne Diseases | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Dose of 200mg doxycycline (Experimental): Treatment of a single dose of 200mg doxycycline
  Interventions: Drug: administration of single dose of doxycycline
- Standard treatment of 5 days doxycycline (200mg at 1st day followed by 4 days of 100mg) (No Intervention): Treatment of 5 days doxycycline (200mg at 1st day followed by 4 days of 100mg)

INTERVENTIONS:
Drug: administration of single dose of doxycycline — Postexposure prophylaxis with Single Dose doxycycline
  Arms: Single Dose of 200mg doxycycline

SUMMARY:
The goal of this clinical trial is to compare standard treatment (5 days of doxycycline) vs single dose doxycycline for the prevention of tick-borne relapsing fever in soldiers who found bite marks on their bodies after an activity that includes contact with the ground or staying at a site suspected of being infected with ticks. The main question[s] it aims to answer are:

* Testing whether preventive treatment with a single dose of doxylin at a dose of 200 mg is effective in preventing recurrent fever, and if so, at what rate
* Checking the profile and rate of side effects in each one of the proposed treatment protocols Participants will be treated with standard treatment (5 days of doxycycline) or single dose doxycycline.

DETAILED DESCRIPTION:
1. In accordance with the guidelines of the Institutional Review Board (IRB), following the completion of the field exercise series, all participating soldiers, both those who actively engaged in the experiment and those who did not, will undergo examination for signs of insect bites.
2. After the medical examination, a treating physician (who is not one of the researchers involved in the study) will determine whether there are signs requiring doxycycline antibiotic treatment for soldiers who participated in the field exercise (regardless of their participation in the research). According to the IRB and IRB guidelines, an Air Force pilot cadet will receive antibiotic treatment if any of the following conditions exist on their body: insect bites, suspicious bites resembling tick bites, or similar symptoms on the spouse of the participant in the exercise.
3. Prophylactic treatment following exposure, whether following a standard doxycycline protocol or a single-dose experimental treatment of 200 mg with a placebo pill, will be administered with instructions on how to take the medication to minimize the risk of side effects, particularly pill esophagitis ("take the medication with plenty of water and remain upright (standing/sitting) for at least half an hour after taking the pill").
4. In cases where it is determined that there is no need for prophylactic treatment, participants will be monitored as an observational control group, distinct from the two experimental arms. In cases where it is decided that treatment is warranted, different approaches will be taken depending on whether the participant is involved in the experiment or not:

   * Non-participating Air Force pilots cadets will be treated according to the standard doxycycline protocol as per IRB guidelines. They will receive doxycycline from the medical facility as prescribed by a physician.
   * Air Force pilots cadets participating in the experiment who are recommended or whose spouses are recommended to receive treatment will receive a packet of pills containing the standard dosage or the experimental treatment, depending on randomization that will occur prior to the distribution of treatment packets. These packets will be provided in advance by the Medical Corps and will be labeled differently according to the dosage. Specifically, a packet containing 6 doxycycline pills at a dosage of 100 mg will be labeled differently from a packet containing 6 pills, with only 2 of them being 100 mg doxycycline, and the rest being placebos. The first two pills containing the active drug will be labeled separately. Only Dr. Yoni Yosef, one of the researcher, will have access to information indicating which label represents the standard dosage and which label represents the experimental dosage. In other words, the physician who examines the soldier and other researchers and study participants will not be exposed to information about which treatment arm the soldier was assigned to, in order to maintain double-blinding. Consequently, a Case Report Form (CRF) documenting the medical examination, treatment decision, and explanation that the soldier participated in the experiment and received either standard doxycycline treatment or a single-dose combination with placebo will be generated.

   Additionally, if a soldier develops a fever within two weeks after participating in the field exercise, it may be indicative of a relapsing fever that was partially treated. In such cases, the soldier will be referred to the Ichilov medical center emergency department for evaluation, with coordination with the principal investigator or the study coordinator, in an organized manner. Furthermore, medical oversight by the Medical Corps' specialist will be provided in cases where an Air Force pilot cadets who did not show any signs of insect bites, but based on a physician's assessment, it is decided that their spouse should receive treatment. This oversight is not dependent on the participation of the Air Force pilot cadets or their spouse in the field exercise or the type of treatment given.
5. Three weeks after the completion of the field exercise series, all participants who attended the field exercise and agreed to participate in the experiment will undergo clinical follow-up, irrespective of whether they required antibiotic treatment. Those not requiring antibiotic treatment will be assessed by a medical officer regarding their medical condition, including signs of relapsing fever and fever. Those who required antibiotic treatment will also be assessed by a medical officer, including an evaluation of signs of relapsing fever, fever, their response to treatment, and follow-up questions regarding the administration of treatment. At this stage, participants in the study, as well as the physicians treating them, will not be aware of which treatment arm they belong to.

   Should participants develop symptoms consistent with relapsing fever or exhibit suspicion of this condition, they will be referred to a medical evaluation in the Ichilov medical center emergency department, in coordination with the principal investigator and the study coordinator. There, blood tests will be conducted, including thick smear for the diagnosis of relapsing fever, along with additional tests as necessary and at the discretion of the hospital physician. The principal investigator will be responsible for referring the soldier to Malram for evaluation, with coordination with the senior hospital epidemiologist.
6. Three weeks after the completion of the field exercise series and the decision regarding treatment, participants in the experiment will complete a digital survey. This survey will be sent to their personal phones to assess side effects of medical treatment or the presence of suspicious symptoms of relapsing fever that were not reported to the medical facility and were not mentioned during the private interview one week after the end of the series. The survey will be filled out using the Microsoft Forms platform, with participant identification based on a serial number provided at the time of informed consent. In other words, there will be no documentation of ID numbers or other identifying information in the generated digital file. The survey will be completed using an online platform such as google or microsoft forms, with participant identification based on a serial number provided at the time of informed consent. Again, there will be no documentation of ID numbers or other identifying information in the generated digital file.
7. Upon completion of the digital survey by all participants of the experiment, the envelopes will be opened, and the researchers will update the electronic medical record with the specific treatment arm to which the participants belonged. Additionally, the study coordinator will inform the battalion's physician in a personalized manner.
8. Each series will be independent of the others, and the same process will be conducted for both series. Prior to each series, participants will sign an informed consent form, and a detailed explanation of all stages will be provided.

Regenerate

ELIGIBILITY:
Inclusion Criteria:

Israel Air Force flight course cadets.

Exclusion Criteria:

* Known sensitivity or allergy to doxycycline
* Fever in the three weeks preceding the performance of the field series
* Suspicion of the Tick borne disease with recurrent fever three weeks before performing the
* Incompletion of the field series

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 526 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Preventing Tick borne recurrent fever | From enrollment to the end of treatment and follow up at 3 weeks
  Examining whether preventive treatment with a single dose of doxycycline at a dose of 200 mg is effective in preventing Tick borne recurrent fever compared to treatment with the standard protocol lasting 5 days

SECONDARY OUTCOMES:
Side effects | From enrollment to the end of treatment and follow up at 3 weeks
  Checking the profile and rate of side effects in each one of the proposed treatment protocols

CONTACTS AND LOCATIONS:
Overall Officials: Barak Gordon, MD, Study Director — Israel defense forces medical corps

IPD SHARING:
Plan to Share IPD: Yes
No individual participant data will be shared. Results will be published by the investigators in academic journals. Sharing of generated study data will be carried out in several different ways. We plan to make our results available to researchers and potential collaborators interested in Tick-borne Relapsing Fever.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 3 months after article publication and the data will be made accessible for up to 96 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact mor.rittblat@mail.huji.ac.il